CLINICAL TRIAL: NCT01145677
Title: Efficacy of Topiramate for Hospitalized Patients With Alcoholism: a 12-Week Randomized, Placebo-Controlled Trial
Brief Title: Efficacy of Topiramate for Hospitalized Patients With Alcoholism
Acronym: ETHoPA-R
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Surinporn Likhitsathian, Department of Psychiatry, Faculty of Medicine, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THoPA-R
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence; Alcoholism; Topiramate
MeSH Terms: conditions — Alcoholism | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topiramate (Experimental)
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — Topiramate 100-300 mg/day orally twice per day
  Other Names: Topamax

SUMMARY:
This is a 12-Week, randomized controlled study of topiramate in hospitalized patients with alcoholism

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized due to alcohol-related problem
* DSM-IV-TR alcohol dependence
* for male: history of alcohol drink >=35/week, female: history of alcohol drink >=28/week for at least 1 week during four weeks prior to the admission
* AUDIT score at least 8
* mild or no alcohol withdrawal symptom
* BMI > 18 kg/m2
* not pregnant and no plan for pregnancy
* intention to decrease or stop drinking

Exclusion Criteria:

* severe psychiatric and cognitive disorders
* other substance dependence, except nicotine and caffeine dependence, during 6 months prior to enrollment
* taking antipsychotics, mood stabilizers, anticonvulsants, opioid analgesics, systemic steroids, carbonic anhydrase inhibitors, hydrochlorthiazide, metformin, pioglitazone, or disulfiram
* unstable medical condition
* medical history of narrow angle glaucoma, renal impairment, kidney stones, and seizures
* moderate to high risk of suicide
* under legal process
* plan to receive a formal treatment for alcoholism from other treatment settings
* pregnancy and nursing woman
* abnormal laboratory tests, including blood urea nitrogen, creatinine, electrolytes, and fasting blood sugar

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Alcohol drink/day | 12 weeks
  Alcohol drink/day assessed by the use of time line follow back

SECONDARY OUTCOMES:
Common adverse effect | 12 week
  Common adverse effect will be assessed by the use of questionaire and self-report

CONTACTS AND LOCATIONS:
Overall Officials: Surinporn Likhitsathian, MD, Principal Investigator — Department of Psychiatry, Faculty of Medicine, Chiang Mai University
Locations (4):
- Thailand (4):
  - Chiang Mai Drug Dependence Treatment Center, Maerim, Chiang Mai
  - Maharaj Nakorn Chiang Mai Hospital, Muang, Chiang Mai
  - Suanprung Psychiatric Hospital, Muang, ChiangMai
  - Maharaj Nakorn Chiang Mai Hospital, Muang, ChiangMai